CLINICAL TRIAL: NCT00676065
Title: Long-term Active Surveillance Study for Oral Contraceptives (LASS)
Status: Completed | Type: Observational
Sponsor: Center for Epidemiology and Health Research, Germany (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Juergen Dinger, MD, PhD, Principal Investigator, Center for Epidemiology and Health Research, Germany
Other Study IDs: ZEG2006_03
Record Dates: First submitted 2008-05-08; First posted 2008-05-12 (Estimated); Results first posted 2014-11-19 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Arterial Thromboembolism; Venous Thromboembolism; Breast Cancer
Keywords: Contraception; Thromboembolism; Breast Cancer
MeSH Terms: conditions — Venous Thromboembolism; Breast Neoplasms; Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: Women who take oral contraceptives containing drospirenone
- 2: Women who take oral contraceptives containing levonorgestrel
- 3: Women who take oral contraceptives containing other progestogens

SUMMARY:
The objective of this study is to characterize and compare the risks of long-term use of oral contraceptives containing drospirenone and of other established oral contraceptives.

DETAILED DESCRIPTION:
The LASS Study is a large, multinational, prospective, controlled, non-interventional, long-term cohort study that follows a series of cohorts. The cohorts consist of new users (first-ever users, switchers and restarters) of three different groups of oral contraceptives (OCs): OCs containing drospirenone (DRSP), OCs containing levonorgestrel (LNG) and OCs containing other progestogens. A "non-interference" approach is used to provide standardized, comprehensive, reliable information on these groups of OCs under routine medical conditions.

The main clinical outcomes of interest for the long-term follow-up are arterial and venous thromboembolism as well as breast cancer. Regular, active contacts with the cohort members (=active surveillance) provide all necessary information on health-related events or changes in health status.

The study is based on the existing long-term EURAS cohorts who are still in follow-up. LASS succeeds EURAS and prolongs the follow-up period for another five years. Total follow-up time of members of the long-term cohorts will be between 6 and 10 years. By means of annual contacts almost all relevant clinical outcomes will be captured. This will be accomplished by contacting the relevant physicians and by reviewing relevant source documents in the case of relevant clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Women who are prescribed an oral contraceptive and who are new users (first-ever users, switchers or restarters) of the formulation

Exclusion Criteria:

* Women who do not consent to participate in the study

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women attending offices of oral contraceptives prescribing physicians
Sampling Method: Non-Probability Sample
Enrollment: 58303 (Actual)
Dates: Start 2001-02; Primary Completion 2011-03 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Dinger, MD, PhD, Principal Investigator — Center for Epidemiology and Health Research Berlin, Germany
Locations (1):
- Center for Epidemiology and Health Research, Berlin, Germany

REFERENCES:
- [Derived] Dinger J, Mohner S, Heinemann K. Cardiovascular risks associated with the use of drospirenone-containing combined oral contraceptives. Contraception. 2016 May;93(5):378-85. doi: 10.1016/j.contraception.2016.01.012. Epub 2016 Jan 26. PMID 26825258

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In the LASS study, 59,510 women were recruited overall. Of these, 836 participants were excluded due to protocol violation (e.g. patient did not start OC use). Furthermore, 371 patients started treatment with non-oral contraceptives. These patients were followed-up but were not part of the per protocol Population (58,303 patients).
Groups:
- Yasmin: Users of oral contraceptives containing 3 mg DRSP and 30 mcg ethinylestradiol
- OC-LNG: Users of oral contraceptives containing levonorgestrel
- OC-other: Users of oral contraceptives containing other progestogens
Period: Overall Study
Arm/Group | Yasmin | OC-LNG | OC-other
Started | 16534 | 15428 | 26341
Completed | 16534 | 15428 | 26341
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- DRSP/EE: Users of oral contraceptives containing 3 mg DRSP and 30 mcg ethinylestradiol
- Total: Total of all reporting groups
Arm/Group | DRSP/EE | OC-LNG | OC-other | Total
Number analyzed (Participants) | 16534 | 15428 | 26341 | 58303
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.9 (8.1) | 25.1 (8.7) | 24.8 (7.8) | 25.2 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16534 | 15428 | 26341 | 58303
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — This study was conducted in seven European countries: Austria, Belgium, Denmark, France, Germany, the Netherlands, and UK.
  participants
    Europe | 16534 | 15428 | 26341 | 58303

OUTCOME MEASURES:

1. Primary Outcome: Arterial Thromboembolism
Description: Arterial thromboembolism associated with the use of oral contraceptives containing drospirenone or levonorgestrel or other progestogens.
Time Frame: Within 10 years
Population: The number of participants refers to the ITT study population. During the course od the study, women could for example stop use of oral contraception at any point of time. Therefore, the woman-years of exposure for each group are provided in addition.
Measure: Number; unit: participants
Units Other Than Participants: Woman-years, AT-population
Arm/Group | DRSP/EE | OC-LNG | OC-other
Number analyzed (Participants) | 16534 | 15428 | 26341
Number analyzed (Woman-years, AT-population) | 52278 | 57539 | 106221
participants | 7 | 22 | 34
Statistical Analysis 1: Comparison: DRSP/EE vs OC-LNG; Tested null hypotheses: the ATE hazard ratio for DRSP/E2 vs. OCs containing LNG is higher or equal to 2; Test type: Non-Inferiority or Equivalence — The LASS study was designed to analyse rare events (incidence rate <1 per 1,000 woman-years and ≥ 1 per 10,000 WY). 300,000 WY of observation would be sufficient to exclude a two-fold risk of rare events in users of DRSP compared to other oral contraceptives with a power (1-β) of 0.80 and an one-sided α of 0.05; Hazard Ratio (HR) = 0.4, 95% CI 2-sided [0.2 to 0.9] — Hazard ratio was adjusted for age, BMI, smoking, hypertension and family history
Statistical Analysis 2: Comparison: DRSP/EE vs OC-other; Tested null hypotheses: the ATE hazard ratio for DRSP/E2 vs. OCs containing other progestogens is higher or equal to 2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.4, 95% CI 2-sided [0.2 to 0.9] — Hazard ratio was adjusted for age, BMI, smoking, hypertension and family history

2. Primary Outcome: Venous Thromboembolism
Description: Venous thromboembolism associated with the use of oral contraceptives containing drospirenone or levonorgestrel or other progestogens.
Time Frame: Within 10 years
Population: as for outcome 1
Measure: Number; unit: participants
Units Other Than Participants: Woman-years, AT population
Arm/Group | DRSP/EE | OC-LNG | OC-other
Number analyzed (Participants) | 16534 | 15428 | 26341
Number analyzed (Woman-years, AT population) | 52278 | 57539 | 106221
participants | 56 | 53 | 144
Statistical Analysis 1: Comparison: DRSP/EE vs OC-LNG; Tested null hypotheses: the VTE hazard ratio for DRSP/E2 vs. OCs containing LNG is higher or equal to 2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.1, 95% CI 2-sided [0.8 to 1.7] — Hazard ratio was adjusted for age, BMI, current duration of use, and family history of VTE
Statistical Analysis 2: Comparison: DRSP/EE vs OC-other; Tested null hypotheses: the VTE hazard ratio for DRSP/E2 vs. OCs containing other progestogens is higher or equal to 2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.7, 95% CI 2-sided [0.5 to 1.0] — Hazard ratio was adjusted for age, BMI, current duration of use, and family history of VTE

3. Primary Outcome: Breast Cancer
Description: Breast cancer associated with the use of hormonal contraceptives either containing both drospirenone (DRSP) and ethinylestradiol (EE), levonorgestrel (LNG) or any other hormonal contraceptive without DRSP.
Time Frame: Within 10 years
Population: as for outcome 1
Measure: Number; unit: participants
Units Other Than Participants: Woman-years
Arm/Group | DRSP/EE | OC-LNG | OC-other
Number analyzed (Participants) | 16534 | 15428 | 26341
Number analyzed (Woman-years) | 52278 | 57539 | 106221
participants | 27 | 31 | 45
Statistical Analysis 1: Comparison: DRSP/EE vs OC-LNG; Tested null hypotheses: the breast cancer hazard ratio for DRSP/E2 vs. OCs containing LNG is higher or equal to 2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.9, 95% CI 2-sided [0.5 to 1.4] — Hazard ratio was adjusted for age, BMI, smoking, educational level and age at menarche
Statistical Analysis 2: Comparison: DRSP/EE vs OC-other; Tested null hypotheses: the breast cancer hazard ratio for DRSP/E2 vs. OCs containing other progestogens is higher or equal to 2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.0, 95% CI 2-sided [0.6 to 1.5] — Hazard ratio was adjusted for age, BMI, smoking, educational level and age at menarche

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected over a time period of 10 years.
Description: ITT population. All study participants were asked for adverse events at each follow-up.
Arm/Group | DRSP/EE | OC-LNG | OC-other
Serious Adverse Events (participants affected / at risk) | 1912/16534 | 2121/15428 | 3936/26341
Other Adverse Events (participants affected / at risk) | 0/16534 | 0/15428 | 0/26341
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DRSP/EE (N=16534) | OC-LNG (N=15428) | OC-other (N=26341)
Infectious diseases (Infections and infestations) | 86 | 86 | 171
Neoplasms, malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 59 | 72 | 124
Neoplasms, benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 96 | 97 | 179
Diseases of the blood and the bloodforming organs (Blood and lymphatic system disorders) | 7 | 9 | 18
Endocrine diseases (Endocrine disorders) | 50 | 74 | 96
Psychiatric & neurological disorders (Psychiatric disorders) | 114 | 136 | 274
Eye (Eye disorders) | 19 | 24 | 40
Ear (Ear and labyrinth disorders) | 24 | 28 | 53
Cardiovascular system (Cardiac disorders) | 198 | 226 | 425
Respiratory system (Respiratory, thoracic and mediastinal disorders) | 56 | 64 | 128
Digestive system (Gastrointestinal disorders) | 248 | 265 | 503
Skin (Skin and subcutaneous tissue disorders) | 82 | 97 | 200
Muscoskeletal system & connective tissue (Musculoskeletal and connective tissue disorders) | 206 | 233 | 403
Genitourinary system (Reproductive system and breast disorders) | 279 | 290 | 572
Pregnancy, delivery & puerperium (Pregnancy, puerperium and perinatal conditions) | 51 | 62 | 99 — SAEs that occurred within 3 months after stop of OC use, were attributed to the last hormonal contraceptive used by the women. Therefore, pregnancy related SAEs on OC cohorts do not necessarily reflect unwanted pregnancies during HC use
Injury, poisoning, accidents, etc. (Injury, poisoning and procedural complications) | 337 | 358 | 651

LIMITATIONS AND CAVEATS:
In non-experimental studies the possibility of bias and residual confounding can never be entirely eliminated. The findings may exclude large, but not small relative risks.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes